CLINICAL TRIAL: NCT03714503
Title: Head Positioning Duration After Retinal Detachment Repair With Vitrectomy and Gas
Brief Title: Head Positioning After Retina Detachment Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00142574
Record Dates: First submitted 2018-10-04; First posted 2018-10-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Retina; Detachment, Rhegmatogenous

STUDY DESIGN:
Intervention Model Description: Simon's two stage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- One day post-operative head positioning (Other): patients will be assigned to remain a one-day post operative head positioning following retina re-attachment surgery
  Interventions: Device: Retina re-attachment repair using C3F8 gas tamponade

INTERVENTIONS:
Device: Retina re-attachment repair using C3F8 gas tamponade — Assigning a one day post-operative head positioning
  Other Names: pars plana vitrectomy

SUMMARY:
This study aims to determine if one day post-operative prone head positioning can be as good as seven days post-operative prone head positioning in patients with retinal detachments with inferior retinal breaks after pars that pars plana vitrectomy (PPV) using perfluoropropane (C3F8) gas as a tamponade. The investigator will conduct a single arm phase II study using a Simon's two-stage design

DETAILED DESCRIPTION:
A. Study Objectives: To determine if one day post-operative prone head positioning can be as good as seven days post-operative prone head positioning in patients with retinal detachments with inferior retinal breaks after PPV using C3F8 gas as a tamponade.

* Primary outcome: retina anatomical success at 3 months post-operatively
* Secondary outcome: retina anatomical success at 1 year post-operatively

B. Study Type and Design: Single arm phase II study to assess its effectiveness and warrant interest in further development. A Simon's two-stage design will be used to test the following hypotheses: null hypothesis (HO): P<=0.6 versus alternative hypothesis (HI): p >= 0.85.

C. Sample size, statistical methods, and power calculation

1. The sample size calculations are based on a Simon's two-stage minimax design. The Investigators plan to recruit 20 patients (20 eyes) with one day post-operative head positioning. This trial will run as a single-arm study in two stages. In the first stage, the Investigators will define a futility rate of 60%. Thus, 11 patients will be enrolled in this stage and if seven or less than seven patients are not declared a "success", the Investigators will terminate this trial after the first stage. If eight or more successes are found in the first stage, the Investigators will continue to the second stage where the Investigators will enroll an additional 9 patients taking the total sample size to 20 patients. The treatment will be considered as promising for future research if the results find that 16 or more than 16 of the 20 patients are declared a 'success' (based on the literature review and a retrospective study, a success rate of 85% is chosen). This minimax design has an expected sample size of 14 patients and a probability of early termination (PET) of 70%. An analogous calculation for the Optimal Simon's design gives a total sample size of 28 but with the same expected sample size of 14, and so the Investigators have decided to adopt the minimax design.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent
* Subjects must be diagnosed with primary rhegmatogenous retinal detachment with inferior breaks
* Subjects must be 18 years and older.
* Women of child-bearing potential must agree to take rapid urine pregnancy test before surgical procedure and have negative result.

Exclusion Criteria:

* pediatric population
* pregnant women
* a previous retinal detachment repair in the study eye
* history of scleral buckling in the study eye
* trauma as a cause of the retinal detachment
* asymptomatic longstanding retinal detachments
* non-compliance with post-operative treatment
* phakic retinal detachment
* exudative retinal detachment
* retinoschisis related retinal detachment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Retina attachment on clinical exam using the indirect ophthalmoscope | 3 months
  Retina remained attached on indirect ophthalmoscopy exam with scleral depression 360 degrees

SECONDARY OUTCOMES:
Retina attachment on clinical exam using the indirect ophthalmoscope | 1 year
  Retina remained attached on indirect ophthalmoscopy exam with scleral depression 360 degrees

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Prairie Village, Kansas, United States

IPD SHARING:
Plan to Share IPD: No